CLINICAL TRIAL: NCT04211935
Title: The Use of Video-assisted Intercostal Nerve Cryoablation, Erector Spinae Block, and Thoracic Epidural for Postoperative Analgesia After Minimally Invasive Repair of Pectus Excavatum
Brief Title: Identification of Best Postoperative Analgesia Method Following a Minimally Invasive Repair of Pectus Excavatum
Acronym: (MIRPE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-2794
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Pectus Excavatum; Pain, Postoperative
MeSH Terms: conditions — Funnel Chest; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomly assigned to one of three interventional groups. Study participants and team members will be blinded on randomized group until entering the operating room, at which point the cryoablation machine and instruments will be brought into the room for INC or the anesthesiologist will place ESB. The PCA pump will be connected to the patient's intravenous line at the end of the case.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Patient Controlled Analgesia (Experimental): This technique involves connecting a patient controlled analgesia pump to the intravenous line. The patient has the ability to push a button to obtain a predetermined dose of an intravenous opioid with a set lockout time period to minimize the potential for over sedation. PCA pumps will be connected to the intravenous line of the patient at the end of the MIRPE operation. anesthesiologists with experience in regional anesthesia.
  Interventions: Device: Use of PCA
- Erector Spinae Block (Experimental): This method consists of the anesthesiologist placing two catheters on each side of the vertebrae which then delivers pain medicine continuously via pumps for 2-3 days post-surgery.
  Interventions: Device: Use of ESB for postoperative pain control after MIRPE
- Intercostal Nerve Cryoablation (Experimental): The INC technique relies on multilevel freezing of the intercostal neurovascular bundle intraoperatively to block sensation and pain for approximately 2 months postoperatively. Trained pediatric surgeons will perform the INC at the time of a MIRPE procedure.
  Interventions: Device: Use of INC for postoperative pain control after MIRPE

INTERVENTIONS:
Device: Use of PCA — A commercially available PCA pump will be connected to the patient's intravenous line at the end of the MIRPE operation.
  Arms: Patient Controlled Analgesia
Device: Use of ESB for postoperative pain control after MIRPE — Pediatric anesthesiologists will place ESB at the time of the MIRPE operation if study participants are randomized into this group.
  Arms: Erector Spinae Block
Device: Use of INC for postoperative pain control after MIRPE — Pediatric surgeons will perform INC during the MIRPE operation if they are randomized to this group.
  Arms: Intercostal Nerve Cryoablation

SUMMARY:
Pectus excavatum is the most common chest wall deformity in children, accounting for 90% of all congenital chest wall deformities. It occurs in one to eight per 1000 live births. The severity of the pectus deformity may become more noticeable during pubertal growth spurs and repair is therefore usually performed in the teenage years. A common operative procedure to repair a pectus deformity is the minimally invasive repair of pectus excavatum (MIRPE). The MIRPE involves the substernal placement of a contoured metal bar secured to the lateral aspect of the ribs. This metal bar allows for correction of the concave deformity by applying constant outward pressure to the underside of the sternum. Although the cosmetic results are excellent, patients do report significant pain from the constant pressure exerted on the chest wall from the metal bar. Pain management approaches tend to differ on both the provider and institutional level. There is a lack of evidence regarding which postoperative analgesia method is best. To address this research gap, this proposal aims to conduct a randomized controlled trail using the three most commonly used methods; 1) patient controlled analgesia (PCA); 2) erector spinae blocks (ESB) with continuous infusion pumps; and 3) video-assisted intercostal nerve cryoablation (INC).

DETAILED DESCRIPTION:
Pectus excavatum deformity is a common condition in a pediatric surgical practice. While MIRPE provides excellent cosmetic results and is associated with shorter operative time and lower intraoperative blood loss, the immediate correction of the concave deformity with a metal bar places patients in a difficult pain control situation. While multiple postoperative analgesia modalities have been studied, there is still a need for a large, prospective, randomized trial that is appropriately powered to evaluate the best pain control modality after MIRPE. Of the clinically appropriate interventions, ESB and INC have been shown to have comparable LOS after the operation, especially when employed as part of an enhanced recovery pathway (ERP) bundle. Comparing these newer analgesia modalities to the more established PCA approach may help identify the most effective postoperative pain control approach that maximizes the safety profile while minimizing the use of narcotic pain medications after MIRPE.

The investigators propose a prospective randomized trial evaluating the effectiveness of INC, PCA and ESB with continuous local anesthetic infusion via a pain pump delivery system. All groups will follow a multimodal enhanced recovery pathway. Groups will different only in the use of INC, PCA, or ESB.

Since previous studies have reported similarly short LOS for both ESB and INC, but no prospective, direct comparisons of these techniques have been done, we believe comparing these two groups to the more established PCA modality will further advance the field of post MIRPE pain management by providing precise estimates of length of stay (LOS), hospital resource utilization, and other important outcomes that have not received sufficient attention including pain, quality of life, resumption of activities of daily living, and a rigorous survey for potential adverse outcomes. The investigators specifically hypothesize that because of the long-term analgesia of up to 2-3 months, the INC group may experience not only shorter LOS but decreased narcotic use than the ESB and PCA groups, and also improved quality of life, with fewer encounters in the postoperative period (30 days) for pain related concerns.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a pectus excavatum deformity that will undergo a MIRPE procedure will be included in the study.

Exclusion Criteria:

* < 13 years old
* > 18 years old
* chronic narcotic preoperative use
* previous repair of pectus excavatum deformity
* previous thoracic surgery
* pregnancy

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 158 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | 24 months
  The investigators will measure the total length of stay following the operation until discharge from the hospital.

SECONDARY OUTCOMES:
Total intravenous and oral opioid use | 24 months
  The investigators will quantify the total opioid usage during the hospitalization and also at home and will convert the total results to morphine equivalences for standardization.
Postoperative pain | 24 months
  The investigators will use reported pain scores to quantify this measure. Scale of 0-10 (0=no pain, 10=worst pain experienced). The investigators will also ask about chest numbness for those in the INC group and will report it on a 0-100% scale (0%=no numbness at all, 100%=completely numb or absent of any sensation).
Quality of life after MIRPE | 24 months
  The investigators will use a questionnaire to identify if patients are back to baseline and performing their activities of daily living. The investigators will also ask about resumption of any sports related activities after the appropriate postoperative restriction timeframe has passed. This will be a multiple choice questionnaire that will record if 1) they are back to baseline, 2) they are almost back to baseline, 3) they are not back to baseline at all. The investigators will also ask in a multiple choice manner if they have resumed their activities of daily living. The possible answers will be 1) Yes, 2) Incorporating some of the preoperative activities, 3) No
Complications | 24 months
  The investigators will ask patients about postoperative complications when they are at home. We will also refer back to the chart for any complications that occur during the initial postoperative period or those that have required a readmission after the initial operation.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Corbitt, MD, Study Director — Safety Officer--University of Texas Southwestern
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No